CLINICAL TRIAL: NCT05433688
Title: Prospective, Mono-center, Randomized, Single-blinded, Controlled Study on the Performance of Symmcora® Mid-term Suture Versus Novosyn® Suture in Patients Undergoing Robotic Assisted Gastric Bypass Surgery
Brief Title: Study on the Performance of Symmcora® Mid-term Suture Versus Novosyn® Suture in Patients Undergoing Robotic Assisted Gastric Bypass Surgery
Acronym: BARGASTRO
Status: Active, not recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1932
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Adiposity
Keywords: gastro-jejunal anastomosis; jejuno-jejunal anastomosis; robotic assisted gastric bypass surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UBS: unidirectional barbed suture (Symmcora® mid term, UBS)
  Interventions: Device: Robotic assisted gastric bypass surgery
- CS: conventional suture (Novosyn®, CS)
  Interventions: Device: Robotic assisted gastric bypass surgery

INTERVENTIONS:
Device: Robotic assisted gastric bypass surgery — The product under investigation and the conventional suture material will be used in routine clinical practice and according to the Instructions for Use (IfU).

SUMMARY:
The study is designed as a prospective, mono-centric, randomized, patient blinded comparison of unidirectional barbed suture (Symmcora® mid term, UBS) vs. a conventional suture (Novosyn®, CS). Patient will be randomly allocated in a 1:1 ratio to either the UBS group or the CS group to perform the gastro-jejunal anastomosis (GJA) and the jejuno-jejunal anastomosis (JJA).

The product under investigation and the conventional suture material will be used in routine clinical practice and according to the Instructions for Use (IfU).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing an elective, primary robotic, assisted gastric bypass surgery (with a BMI ≥40 kg/m2 or with a BMI ≥35 kg/m2) with one or more of the following comorbidities: refractory arterial hypertension, type 2 diabetes mellitus and/or proven sleep apnea) with the need to close the gastro-jejunal anastomosis (GJA) and jejuno-jejunal anastomosis (JJA).
* Age ≥18 years
* Written informed consent

Exclusion Criteria:

* Emergency surgery
* Previous gastric surgery
* History of chronic steroid use
* Pregnancy or breastfeeding
* Patients with hypersensitivity or allergy to the suture material
* Non compliance
* Participation in another randomized controlled trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective primary, robotic assisted gastric bypass surgery with the need to close the gastro-jejunal anastomosis and the jejuno-jejunal anastomosis.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Time to perform the anastomosis | intraoperatively
  Time to perform the gastro-jejunal anastomosis and the jejuno-jejunal anastomosis

SECONDARY OUTCOMES:
Anastomotic leak rate over postoperative period | until discharge (approximately 10 days after surgery), at 30 days and at 12 months postoperatively
  Number of patients having Anastomotic leak at each examination
Anastomosis stenosis rate over postoperative period | until discharge (approximately 10 days after surgery), at 30 days and at 12 months postoperatively
  Number of patients having Anastomosis stenosis at each examination
Gastric fistula rate over postoperative period | until discharge (approximately 10 days after surgery), at 30 days and at 12 months postoperatively
  Number of patients having Gastric fistula at each examination
Rate of Obstruction over postoperative period | until discharge (approximately 10 days after surgery), at 30 days and at 12 months postoperatively
  Number of patients having obstruction of the anastomosis at each examination
Rate of Anastomosis bleeding over postoperative period | until discharge (approximately 10 days after surgery), at 30 days and at 12 months postoperatively
  Number of patients having anastomosis bleeding at each examination
Cumulative Frequency of other complications according to "Clavien-Dindo" over postoperative period | until discharge (approximately 10 days after surgery), at 30 days and at 12 months postoperatively
  Number of other complications classified according to "Clavien-Dindo" classification in order to rank a complication in an objective and reproducible manner. It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). The introduction of the subclasses a and b allows a contraction of the classification into 5 grades (I, II, III, IV and V) depending on the size of the population observed or the of the focus of a study. Complications that have the potential for long-lasting disability after patient's discharge (e.g.: paralysis of a voice cord after thyroid surgery) are highlighted in the present classification by a suffix ("d" for disability). This suffix indicates that a follow-up is required to comprehensively evaluate the outcome and related long-term quality of life
Rate of Re-anastomosis over postoperative period | until discharge (approximately 10 days after surgery), at 30 days and at 12 months postoperatively
  Number of re-anastomosis at each examination
Total operation duration | intraoperatively
  time from cut to closure in minutes. The time is rounded up and only whole numbers are used
Total procedure costs | until discharge approximately 10 days after surgery
  Costs (15 Euro / Operation minute; suture material, number of used sutures, costs / Hospital day)
Length of postoperative stay | until discharge approximately 10 days after surgery
  Number of days after surgery until the patient is discharged from hospital
Patient satisfaction (VAS) | until discharge (approximately 10 days after surgery), at 30 days and at 12 months postoperatively
  With the Visual Analogue Scale from 0 mm - 100 mm the satisfaction of the patient will be evaluated with 0 (not satisfied at all) to 100 (very satisfied).
Patient pain (VAS) | until discharge (approximately 10 days after surgery), at 30 days and at 12 months postoperatively
  With the Visual Analogue Scale from 0 mm - 100 mm the pain of the patient will be evaluated with 0 (no pain) to 100 (worst pain).
Bariatric Analysis and Reporting Outcome System (BAROS) | preoperative, 30 days and 12 months post-surgery
  questionnaire a common tool to evaluate patient's outcome and quality of life before and after bariatric surgeries. Three main parameters are evaluated with this tool, the weight, the medical conditions and the quality of life. The weight and the medical conditions will be evaluated by the physician. The questions regarding the quality of life will be answered directly by the patients. The six categories (felling, sexual activities, physical activities, work, food and social contacts) can be answered on scale with 10 steps from very good to very bad.
Course of Health Status measured with EQ-5D-5L Score | preoperative, 30 days and 12 months post-surgery
  EQ-5D-5L is a Quality of Life Score introduced by the EuroQol Group. The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  Descriptive system comprises five dimensions (5D): mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension has 5 levels (5L): no problems, slight problems, moderate problems, severe problems, extreme problems. Each answer results in a 1-digit number. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Assessment of the handling of the unidirectional barbed suture | intraoperatively
  intra-operatively including different dimensions with 5 evaluations levels (excellent, very good, good, satisfied, poor).
Assessment of the barbed suture compared to a conventional suture | intraoperatively
  Handling of barbed suture compared to a conventional suture (degree of difficulties and ease of handling) measured in two categories with a 5 point scale (strongly disagree, disagree, neither agree nor disagree, agree, strongly agree)

CONTACTS AND LOCATIONS:
Overall Officials: Jan H Beckmann, Dr., Principal Investigator — University Hospital Schleswig-Holstein
Locations (1):
- Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beckmann JH, Baumann P, Jackisch C, Richter F, Mehdorn AS, Becker T, Taivankhuu T, von Schonfels W. Assessment of a new unidirectional barbed suture versus a conventional suture for anastomosis during robotic-assisted Roux-en-Y gastric bypass surgery in obese patients: BARGASTRO - study protocol for a German randomized active-controlled trial. Trials. 2026 Jan 6;27(1):87. doi: 10.1186/s13063-025-09401-9. PMID 41495768